CLINICAL TRIAL: NCT07225491
Title: A Prospective Registry of Patients Undergoing Surgical Decompression Followed by Radiation Therapy for Spine Tumors
Brief Title: Spine Oncology Registry
Status: Recruiting | Type: Observational
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: Icotec Medical, Inc (Unknown)
Responsible Party: Principal Investigator, James Elder, Principal Investigator, Ohio State University Comprehensive Cancer Center
Other Study IDs: 20253216; NCI-2024-07629 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); OSU-23207 (Other: Ohio State University Comprehensive Cancer Center)
Record Dates: First submitted 2025-10-14; First posted 2025-11-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Spine Tumor; Spine Metastases; Spine Cancer
MeSH Terms: conditions — Spinal Cord Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study to evaluate hardware related and oncologic outcomes in adult patients with primary and metastatic spine disease undergoing separation surgery followed by radiation treatment.

DETAILED DESCRIPTION:
This study is being done to collect information about patients undergoing separation surgery followed by radiation for the treatment of primary and metastatic spine disease. Participants will be asked to complete some patient reported outcome questionnaires and researchers will collect information from medical records to evaluate oncologic and hardware related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary or metastatic disease to the spine who undergo surgical decompression and stabilization followed by radiation therapy

Exclusion Criteria:

* Inability to obtain a standard MRI or CT / CT myelogram for radiation treatment planning and dosimetry
* Inability to receive radiation treatment.
* Patients under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be comprised of patients with primary and metastatic spine disease who undergo surgery followed by radiation therapy.
  Patients may be enrolled regardless of previous local or systemic treatments received prior to enrollment in this registry.
  Patients may be enrolled regardless of other current local or systemic treatments of disease extent.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12, 18, 24 months
Local control of treated lesion based on radiographic review | 3, 6, 9, 12, 15, 16, 21, 24 months
  Patients will be classified as achieving local control if demonstrating response of treated spine lesion after treatment. Local control will be assessed by comparing the radiographic images after treatment and prospectively every 3 months for up to 24 months
Progression free survival | 3, 6, 9, 12, 15, 16, 21, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James B Elder, MD, Principal Investigator — Ohio State University
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers Robert wood Johnson Medical School, New Brunswick, New Jersey
  - The Ohio State University Wexner Medical Center, Columbus, Ohio